CLINICAL TRIAL: NCT06763198
Title: Genetic Polymorphisms Associated With the Risk of Pancreatitis in Patients With Alcohol Related Cirrhosis.
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Cirrhosis-71
Record Dates: First submitted 2025-01-01; First posted 2025-01-08 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Alcohol-related Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alcohol-related cirrhosis: Alcohol-related cirrhosis
- Liver cirrhosis of other etiologies: Liver cirrhosis of other etiologies

SUMMARY:
Alcohol is a known risk factor for both pancreatitis and cirrhosis. However, not all patients with alcohol related cirrhosis develop pancreatitis. It is not known which patients with alcohol-related cirrhosis develop symptomatic or clinically inapparent pancreatitis (Acute or Chronic Pancreatitis).There is no data whether genetic polymorphisms predispose patients with alcohol-related cirrhosis to additional pancreatic injury. There is no data on the spectrum of clinical and subclinical pancreatic changes (structural and functional) in patients with alcohol-related cirrhosis, and their genotypic correlates.This study aims to determine pancreatitis-related gene variants among patients with alcohol-related cirrhosis, with and without pancreatitis. We also aim to study differences in nutritional and functional parameters among alcoholic cirrhosis with and without chronic pancreatitis and also define the relationship of genetic polymorphisms with the pancreatic phenotype. Consecutive patients with alcohol related cirrhosis will be screened for changes of pancreatitis on CT/MR/EUS. Those with and without pancreatitis will be compared with respect to demographic, clinical, genotype, nutritional status .We will also be including a group of MAFLD/Cryptogenic cirrhosis for genotypic and phenotypic comparison.

DETAILED DESCRIPTION:
Aim and Objective - To determine pancreatitis-related gene variants among patients with alcohol-related cirrhosis, with and without pancreatitis.

Primary objective: To determine the genetic variants associated with morphological and functional pancreatic changes among patients with alcohol-related cirrhosis.

Secondary objectives

1. To define the relationship of genetic polymorphisms with the pancreatic phenotype.*
2. To study differences in nutritional and functional parameters among alcoholic cirrhosis with and without chronic pancreatitis.

Hypothesis -

- Genetic polymorphisms related to pancreatitis predispose patients with alcohol-related cirrhosis to additional pancreatic injury.

Associated chronic pancreatitis (clinically apparent or subclinical) negatively influences the nutritional and functional status of patients with alcohol-related cirrhosis

* Study design: Cross sectional study of two study cohorts
* Study period: 1 year.
* Sample size with justification: Studies have reported pathogenic SPINK 1 mutations in 25% -50.0% among idiopathic CP and 10-20% in acute pancreatitis as compared to 1%-4.7% among controls. The investigator assume pathogenic SPINK 1 mutation frequency of 50% and 1% among alcohol-related cirrhosis with and without CP, respectively. The investigator also assume a 33% prevalence of CP among alcohol-related cirrhosis. With significance (α) at 0.5, power of 80%, investigator need to enroll 100 patients of alcohol-related cirrhosis.The investigator will also include a cohort of 50 males with cirrhosis of other etiologies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years of age.
2. Alcohol-related cirrhosis
3. Males

Exclusion Criteria:

1. Current Hepatic encephalopathy or cognitive dysfunction precluding adequate nutritional and functional assessment.
2. HCC.
3. Complete or partial PVT.
4. Significant cardio-pulmonary comorbidity
5. Patients who do not consent for genetic study
6. Inability to provide informed consent.
7. Cannot understand Hindi or English should be excluded since they will not be able to reply objectively to questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Study Population: * Patients > 18 years of age.
  * Who have either alcohol related or non alcohol related cirrhosis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-25 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Genetic polymorphisms in one or more pancreatitis-associated genes* among patients with alcohol-related cirrhosis, with and without pancreatitis. | Day 0

SECONDARY OUTCOMES:
Differences in genetic polymorphisms in one or more pancreatitis related genes in patients with pancreatitis between alcohol related cirrhosis and cirrhosis of other etiologies. | Day 0
To define the relationship of genetic polymorphisms with the pancreatic phenotype.* | Day 0
Prevalence of pancreatitis defined by CT/MR/EUS among patients with alcohol-related cirrhosis. | Day 0
Difference in prevalence of pancreatitis defined by CT/MR/EUS among patients with alcohol-related cirrhosis and cirrhosis of other etiologies . | Day 0
Severe exocrine insufficiency defined by fecal elastase <100µg/g stool among cirrhotic patients with and without chronic pancreatitis | Day 0
Endocrine insufficiency defined by FBS >126mg/dl and HbA1c >6.5% among cirrhotic patients with and without chronic pancreatitis. | Day 0
Sarcopenia defined by Skeletal muscle index of < 50cm/m2 in men on CT, and/or 7.0 kg/m2 on DEXA among cirrhotic patients with and without chronic pancreatitis. | Day 0
Liver frailty index > 4.5 | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided